CLINICAL TRIAL: NCT02071641
Title: Phase II Study of Sunitinib Rechallenge in Patients With Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/259
Record Dates: First submitted 2013-09-27; First posted 2014-02-26 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Patients will be treated in repeated 6-week cycles with 50 mg sunitinib orally daily for 4 weeks followed by 2 weeks off.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib

SUMMARY:
Targeted therapies are associated with (acquired) resistance after a median of 5-11 months of treatment, resulting in disease progression, while almost no tumors are intrinsically resistant in the first line setting. The investigators recently published that tumor cell resistance to sunitinib may be directly related to lysosomal sequestration of sunitinib. This resistance mechanism was shown to be transient, since a drug-free culture period could normalize the lysosomal storage capacity for sunitinib and resulted in recovery of drug sensitivity.

In two reports it has been suggested that patients with metastatic Renal Cell Carcinoma who responded to sunitinib in the first-line setting may benefit from rechallenge with sunitinib after failure of second-line treatment. However, these data are retrospective. A prospective trial to investigate a rechallenge with sunitinib is needed to determine whether this strategy is of benefit for patients with mRCC with prior clinical benefit to sunitinib but who stopped treatment because of overt clinical resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed clear-cell mRCC.
2. Patients who progressed on first-line treatment with sunitinib and who had clinical benefit defined as a response (according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria) or SD for more than 6 months on this treatment.
3. Patients who progressed after second-line treatment (mTOR inhibitor or other treatment as long as patients are not treated with a Vascular Endothelial Growth Factor (VEGF) targeted Tyrosine Kinase Inhibitor (TKI), see exclusion criteria), or who progressed after a treatment-free interval of at least 3 months since discontinuation of first-line sunitinib treatment.
4. Patients with radiological (and/or clinical) confirmed progressive disease according to RECIST 1.1 criteria.
5. Measurable or evaluable disease as defined by RECIST 1.1.
6. WHO performance status 0-2.
7. Life expectancy of at least 12 weeks.
8. Age 18 years or older.
9. Able to receive oral medication.
10. Able to provide written informed consent.
11. Adequate hematologic function: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, Hb ≥ 6.0 mmol/L.
12. Patients with brain metastases are eligible if they have been stable for at least two months post-radiation therapy or surgery.
13. No other current malignant disease, except for basal cell carcinoma of the skin.
14. Adequate hepatic function: serum bilirubin ≤ 1.5 x Upper Limit of Normal (ULN), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 x ULN (or ≤ 5 times ULN if liver metastases are present).
15. Renal function: estimated glomerular filtration rate ≥ 40 ml/min.
16. Patients with reproductive potential must use effective contraception. Female patients must have a negative pregnancy test.

Exclusion Criteria:

1. Patients treated with any VEGF targeted TKI (sorafenib, pazopanib, axitinib, dovitinib) as second-line treatment after progression on first-line sunitinib treatment.
2. Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 2 separate measurements on at least 2 separate days.
3. Active infection or serious intercurrent illness.
4. Presence of unstable angina, recent myocardial infarction (within the previous 3 months).
5. Macroscopic hematuria.
6. Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance.
7. Any other major illness that, in the investigator's judgment, substantially increases the risk associated with the subject's participation in the study.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | After 3 months of treatment
  To investigate the proportion of patients with metastic Renal Cell Carcinoma retreated with sunitinib that is progression-free at 3 months.

SECONDARY OUTCOMES:
Clinical benefit rate | progression free at 3 months
  To assess the clinical benefit rate (ORR and SD), median Progression Free Survival (mPFS) and Overall Survival (OS) in individuals retreated with sunitinib.
Effects of sunitinib rechallenge on LAMP1/2 proteins | Blood samples will be collected at baseline, t=4 wk, t=6 wk, t=12 wk and at the end of study treatment (disease progression and/or death)
  To assess the effects of sunitinib rechallenge on Lysosome-associated membrane protein 1/2(LAMP1/2) proteins in Peripheral Blood Mononuclear Cells and tumor tissue.
The immunological effects of sunitinib rechallenge | Blood samples will be collected at baseline, t=4 wk, t=6 wk, t=12 wk and at the end of study treatment (disease progression and/or death).
  To assess the immunological effects of sunitinib rechallenge on the number and activation state of circulating Dendritic Cell(DC), Myeloid-Derived Suppressor cell (MDSC) and Regulatory T-cell (Tregs).
Mass spectrometry-based identification of phosphorylated proteins in tumor tissue during treatment | Blood samples will be collected at baseline, t=4 wk, t=6 wk, t=12 wk and at the end of study treatment (disease progression and/or death).
  To study phosphoproteomic profiles of tumors before rechallenge and at the time of progression. LC-MS/MS-based phospho-proteomics for the identification of sunitinib response and resistance biomarkers
Concentrations of sunitinib | Blood samples will be collected at baseline, t=4 wk, t=6 wk, t=12 wk and at the end of study treatment (disease progression and/or death).
  To assess sunitinib drug levels and tumor tissue concentrations of sunitinib.
Effect of retreatment | progression free at 3 months
  To evaluate the effect of retreatment with sunitinib on the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- VU Medical Center, Amsterdam, Netherlands